CLINICAL TRIAL: NCT00220662
Title: The Efficacy of Readiness and Motivation Therapy in Individuals With Anorexia Nervosa and Bulimia Nervosa
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Paul's Hospital, Canada (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCM99-0177
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2004-07

CONDITIONS: Anorexia Nervosa; Bulimia Nervosa
Keywords: anorexia nervosa; bulimia nervosa; readiness and motivation
MeSH Terms: conditions — Anorexia Nervosa; Bulimia Nervosa

INTERVENTIONS:
Behavioral: Readiness and Motivation Therapy

SUMMARY:
This research examines the efficacy of a 5-session individual psychotherapy intervention designed to enhance readiness and motivation for change in individuals with anorexia nervosa, bulimia nervosa, and eating disorder not otherwise specified.

It is hypothesized that individuals randomly assigned to receive Readiness and Motivation Therapy (RMT) will have higher readiness and motivation scores and improved eating disorder and psychiatric symptomatology following the intervention than individuals assigned to a no-treatment control condition.

DETAILED DESCRIPTION:
Readiness and motivation for change is a significant concern in the treatment of individuals with eating disorders, as evidenced by frequent treatment drop-out, refusal, and relapse. This research examines the efficacy of a 5-session intervention designed to enhance readiness and motivation for change in individuals with anorexia nervosa. A manualized treatment protocol of Readiness and Motivation therapy (RMT) has been developed. It is hypothesized that individuals randomly assigned to RMT will have improved readiness and motivation for change as assessed using the Readiness and Motivation Interview (RMI) at post-treatment, 3-month, and one-year follow-up than individuals assigned to a no treatment control condition. If RMT proves to be effective, it could be added to the menu of treatment options, to permit for better tailoring of treatment to client readiness for change.

ELIGIBILITY:
Inclusion Criteria:

* meet DSM-IV diagnostic criteria for anorexia nervosa, bulimia nervosa, or eating disorder not otherwise specified

Exclusion Criteria:

* acute medical crisis
* acute psychiatric crisis

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100
Dates: Start 2000-06; Study Completion 2006-06

PRIMARY OUTCOMES:
Readiness and Motivation Scores Post-treatment and at 3-month and one-year follow-up

SECONDARY OUTCOMES:
Psychiatric and eating disorder symptom severity Post-treatment and at 3-month and one-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Josie Geller, Ph.D., Principal Investigator — St. Paul's Hospital, Department of Psychiatry/University of British Columbia, Department of Psychiatry
Locations (1):
- Eating Disorders Program, St. Paul's Hospital 1081 Burrard St., Vancouver, British Columbia, Canada